CLINICAL TRIAL: NCT07072377
Title: Nutritional Prehabilitation to Improve Cancer Outcomes (N-PICO)
Acronym: N-PICO
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Vermont Medical Center (Other)
Responsible Party: Principal Investigator, Randall F Holcombe, Director-Faculty, University of Vermont Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UVMCC2501
Record Dates: First submitted 2025-05-22; First posted 2025-07-18 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Malnutrition; Cancer-related Malnutrition; Quality of Life (QOL); Nutritional Support; Nutritional Interventions; Rural Health
Keywords: Cancer Nutrition Intervention; Malnutrition in Cancer Patients; Nutritional Support for Cancer; Prehabilitation Program for Cancer; Rural Cancer Nutrition; Quality of Life and Cancer Nutrition; Remote Nutritional Consultations; Cancer Treatment Outcomes and Nutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Rural, Remote, Low-Intensity (Experimental): Rural, Remote, Low-Intensity
  Interventions: Behavioral: Intensity of Nutritional Intervention
- Rural, Remote, High-Intensity (Experimental): Rural, Remote, High-Intensity
  Interventions: Behavioral: Intensity of Nutritional Intervention
- Urban, Remote, Low-Intensity (Experimental): Urban, Remote, Low-Intensity
  Interventions: Behavioral: Intensity of Nutritional Intervention; Behavioral: Remote or In-Person
- Urban, Remote, High-Intensity (Experimental): Urban, Remote, High-Intensity
  Interventions: Behavioral: Intensity of Nutritional Intervention; Behavioral: Remote or In-Person
- Urban, In-Person, Low-Intensity (Experimental): Urban, In-Person, Low-Intensity
  Interventions: Behavioral: Intensity of Nutritional Intervention; Behavioral: Remote or In-Person
- Urban, In-Person, High-Intensity (Experimental): Urban, In-Person, High-Intensity
  Interventions: Behavioral: Intensity of Nutritional Intervention; Behavioral: Remote or In-Person

INTERVENTIONS:
Behavioral: Intensity of Nutritional Intervention — Participants will either receive High or Low intensity nutritional support.
Behavioral: Remote or In-Person — Patients will either receive their support in-person or remotely.
  Arms: Urban, In-Person, High-Intensity; Urban, In-Person, Low-Intensity; Urban, Remote, High-Intensity; Urban, Remote, Low-Intensity

SUMMARY:
Brief Summary

The goal of this clinical trial is to evaluate the acceptability and adherence of low- and high-intensity remote nutritional interventions for cancer patients in rural and urban areas, specifically focusing on those with invasive cancer who are about to start treatment. The main question[s] it aims to answer are:

Can low- and high-intensity remote nutritional interventions improve adherence to cancer treatment and quality of life? What is the impact of nutritional support on treatment delays, unplanned healthcare utilization, and dietary modifications? Researchers will compare the low-intensity arm (initial nutritional consultation plus written materials) to the high-intensity arm (1-hour consultation, monthly follow-ups, and written materials) to see if higher intensity interventions lead to better outcomes in terms of adherence, quality of life, and healthcare utilization.

Participants will:

Receive either a low- or high-intensity nutritional consultation. Complete surveys assessing quality of life, dietary habits, treatment delays, and unplanned healthcare use.

Be asked to participate in monthly follow-up consultations (for the high-intensity group) to track progress and provide additional support.

DETAILED DESCRIPTION:
This randomized, two-arm pilot study evaluates the feasibility, acceptability, and clinical impact of low- and high-intensity remote nutritional interventions for patients with invasive cancer who are initiating treatment. The study targets both rural and urban populations and will enroll participants at the University of Vermont Cancer Center and affiliated sites across Vermont and northern New York.

Participants are randomly assigned to one of two intervention arms:

Low-Intensity Arm: Participants receive a one-time remote nutritional consultation and a packet of standardized educational materials, designed to provide foundational guidance on protein and calorie intake during cancer treatment.

High-Intensity Arm: Participants receive an initial 1-hour consultation followed by monthly follow-up consultations (total of three across six weeks), in addition to the same educational materials. The goal is to offer personalized and sustained support throughout the course of treatment.

The interventions are delivered remotely to reduce logistical burden and improve accessibility, particularly for patients in rural settings.

The study's primary objective is to evaluate the feasibility of implementing these remote interventions, measured by participant adherence to scheduled consultations and dietary goals. Secondary objectives include assessments of acceptability (via structured participant surveys) and exploratory evaluation of changes in quality of life, dietary behaviors, treatment adherence, and unplanned healthcare utilization.

Validated tools used include the FACT-G (Functional Assessment of Cancer Therapy-General), a brief satisfaction survey, and the NHANES Dietary Screener Questionnaire. Clinical and utilization data (e.g., treatment delays, emergency department visits, unplanned hospitalizations) will be abstracted from the medical record.

This pilot study is intended to inform the design of a future larger trial by generating preliminary data on the practicality and clinical utility of nutritional prehabilitation strategies, especially for underserved cancer patients in rural areas.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of invasive cancer with plans to initiate chemo-, immune-, targeted-, or hormonal therapy for treatment of their malignancy, or within one month of starting treatment.
* Age ≥ 18 years of age.
* Patients must be able to read, write, and speak English as study material and virtual nutrition consultation calls are only available in English.
* Patients receiving treatment at a participating ambulatory medical oncology site.
* Willingness to have a remote nutritional consultation and complete questionnaires/surveys.
* Patients must be informed of the investigational nature of this study and must sign and give written informed consent in accordance with institutional and federal guidelines.

Exclusion Criteria:

* Diagnosis of acute leukemia (these patients generally receive predominantly inpatient care).
* Diagnosis of head & neck cancer, esophageal cancer, gastric cancer, patients presenting with recognized cachexia or severe malnutrition, or patients with PEG tubes for enteral feeding.

Rationale: These patients would normally be referred for dietary consultation and may need ongoing clinical intervention from an on-site dietitian beyond the period of the proposed study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2028-05 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Adherence to Assigned Nutritional Intervention (Low- vs. High-Intensity) | 6 months
  Adherence will be assessed over the 6-week intervention period using two metrics:
  1. Proportion of scheduled dietary counseling contacts completed (≥70% completion threshold), and
  2. Participant self-report of meeting ≥70% of individualized nutrition goals, recorded weekly.
  Adherence will be summarized as the percentage of participants in each arm who meet both criteria.
  Unit of Measure: Percentage of participants meeting adherence threshold (%)
Acceptability of Nutritional Intervention Based on Participant Survey | 6 months
  Acceptability will be measured at the end of the 6-week intervention using a structured participant survey developed for the study. This survey includes Likert-scale questions (e.g., ease of use, satisfaction, perceived helpfulness) and open-ended feedback. Responses will be analyzed to compare acceptability between low- and high-intensity intervention arms.
  Unit of Measure: Mean score on acceptability survey

SECONDARY OUTCOMES:
Change in Quality of Life Measured by the PROMIS Global Health Scale | 6 months
  Participant quality of life will be measured using the PROMIS Global Health v1.2 questionnaire at baseline and after the 6-week intervention. This tool provides T-scores for physical and mental health domains. Changes in mean T-scores will be compared between intervention arms.
  Unit of Measure: Mean change in PROMIS T-scores (range: 0-100; higher scores = better health)
Patient-Reported Dietary Behavior Change | Unit of Measure: Proportion of participants reporting positive dietary change (%)
  Participants will report dietary behavior changes related to protein and calorie intake via a structured questionnaire administered at 6 weeks. Survey results will include frequency of changes (e.g., increased protein intake) and perceived ease of implementation.
Frequency of Treatment Delays or Modifications During Chemoradiation | 6 months
  Treatment delays or dose modifications (e.g., chemotherapy hold, radiation rescheduling) will be extracted from the EMR and documented during the 6-week treatment window.
  Unit of Measure: Number of delays or modifications per participant
Unplanned Healthcare Utilization (ER Visits and Unplanned Hospitalizations) | 6 months
  The number of unplanned emergency room visits and unplanned hospital admissions during the intervention period will be recorded and compared between arms.
  Unit of Measure: Count of ER visits or unplanned hospitalizations per participant

CONTACTS AND LOCATIONS:
Locations (1):
- University of Vermont Medical Center, Burlington, Vermont, United States

IPD SHARING:
Plan to Share IPD: No
Anonymized patient related data will be incorporated into publications and will be made available to other investigators at reasonable request.